CLINICAL TRIAL: NCT06357442
Title: Assessment of Endometrial Thickness Among Adolescent and Young Adult Patients on Estrogen Replacement Therapy Using Continuous Oral Micronized Progesterone Versus the Etonogestrel Implant: a Prospective Pilot Study
Brief Title: Assessment of Endometrial Thickness Among Adolescent and Young Adult Patients on Estrogen Replacement Therapy Using Daily Oral Micronized Progesterone Versus the Etonogestrel Implant.
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 23-2305
Record Dates: First submitted 2024-03-14; First posted 2024-04-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Primary Ovarian Insufficiency; Hypogonadotropic Hypogonadism; Hormone Replacement Therapy
Keywords: hormone replacement therapy; hypogonadism; primary ovarian insufficiency; endometrial protection; progesterone replacement therapy
MeSH Terms: conditions — Primary Ovarian Insufficiency; Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Daily oral micronized progesterone: On estrogen replacement therapy using 100mg oral daily micronized progesterone
- Etonogestrel implant (Nexplanon): On estrogen replacement therapy with etonogestrel implant in place

SUMMARY:
The goal of this observational study is to compare endometrial stripe thickness in adolescent and young adult (AYA) patients with a uterus on estrogen replacement therapy using oral progesterone versus the etonogstrel implant for endometrial protection.

The main questions it aims to answer are:

Aim 1: Characterize the mean endometrial thickness in AYA on estrogen hormone replacement therapy before initiation of progesterone therapy

Aim 2: Characterize the mean changes and variability in endometrial thickness in AYA treated for 6 months with either the etonogestrel implant or continuous oral progesterone

Aim 3: Assess satisfaction, side effects, bleeding patterns, any progesterone modifications, and adherence in AYA treated for 6 months with either etonogestrel implant or continuous progesterone

Participants will be asked to:

* Get two pelvic ultrasounds
* Fill out two surveys
* Continue their current hormone replacement therapy
* Initiate one of two progesterone therapies (prometrium 100mg daily or Nexplanon)

Researchers will compare the change in endometrial thickness after 6 months of progesterone use to see if there is a significant difference in the mean change between the prometrium and Nexplanon groups.

DETAILED DESCRIPTION:
Study Design and Research Methods This study is a prospective, observational pilot study to assess the acceptability of study procedures and describe initial trends in our outcomes of interest, including endometrial stripe thickness among patients on estrogen replacement therapy after six months of either continuous oral micronized progesterone or etonogestrel implant. Participants will self-select into one of two study arms: (1) oral micronized progesterone (Prometrium), 100mg daily; or (2) etonogestrel implant (Nexplanon).

Recruitment and Enrollment Providers will identify eligible patients at routine appointments in the Children's Hospital Colorado Pediatric and Adolescent Gynecology Clinics, Endocrine Clinic, Oncofertility Clinic, and Multidisciplinary Turner Syndrome Clinic. Providers will briefly discuss the study to assess patient interest and, if the patient expresses interest, patients will be approached by a member of the study team for potential study enrollment. A member of the study team will provide an in-depth explanation of the study, answer any questions, and review the informed consent form.

If a patient decides to participate in the study, they or their legal guardian will provide a digital signature on the eConsent form (and eAssent form for participants aged 12-17). If participants would like a copy of the eConsent form, a signed copy will be emailed to the address they provide. The original consent will be stored in the secure, password protected REDCap database.

Feasibility and Timeline We will be enrolling from the following Children's Hospital Colorado-affiliated clinics: Pediatric and Adolescent Gynecology Clinic, Endocrine Clinic, Oncofertility Clinic, and Multidisciplinary Turner's Clinic. Each of these clinics routinely treats pediatric and adolescent patients requiring hormone replacement therapy. We anticipate meeting enrollment goals within one year. In a review of ICD codes for primary ovarian failure, 313 patients presented to CHCO from October 1, 2022 to October 1, 2023. Of these patients, 87 were under the age of 25 and received prescriptions for estradiol. We anticipate a 15% enrollment rate (3-4 patients per month) which translates to an 11-to-12-month enrollment period. We also anticipate that recruitment in the oral progesterone arm will be significantly higher compared to the etonogestrel implant group (~7:1) based on clinical experience. Thus, we anticipate that recruitment may take longer in this group but will not have an enrollment timing estimate until enrollment begins. The recruitment timing of this pilot study will help inform the timeline and feasibility of a full study in the future.

Due to lack of existing literature, we do not know the optimal time to assess changes in endometrial thickness after hormone initiation in this exact study population. ACOG clinical consensus for endometrial hyperplasia is to perform histologic re-assessment of the endometrium 3-6 months after initiating progestin therapy for treatment.27 The initial clinical trials for the etonogestrel implant reference counseling patients that their bleeding pattern after 3-6 months of use will persist due to hormonal influence on the endometrium.24 Additionally, the only available study on the effect of desogstrel (the precursor hormone to etonogestrel) on endometrial protection and menstruation normalization among reproductive aged women was a 6 month randomized control trial. 25 Thus, by extrapolating this available data we will plan on a 6 month study timeline to allow enough time for endometrial changes to occur before performing a repeat ultrasound.

Data Collection The study team will conduct a base-line survey over the phone to collect relevant clinical history (e.g., ovarian failure diagnoses, previous hormone treatments etc.), stored securely in a REDCap database.

Participants will have a formal limited transabdominal pelvic ultrasound performed at two time points during the study. The first ultrasound will be performed at enrollment (baseline) on estrogen therapy alone to measure endometrial thickness prior to initiation or progesterone. Baseline ultrasounds will be ordered and scheduled for the patient at Children's Hospital Colorado at enrollment. Radiology technicians will perform the ultrasound, and a radiologist will confirm and report ultrasound results in the participant's medical record per standard of care.

After a baseline ultrasound is obtained, participants will initiate their selected progesterone therapies. Participants that select to oral progesterone will be prescribed 100mg oral micronized progesterone daily (Prometrium) for 6 months. Participants who elect for an etonogestrel implant will have a clinic appointment made in the Pediatric and Adolescent Gynecology Clinic at Children's Hospital Colorado for a Nexplanon insertion that will be performed per standard protocol. The study team will track the date of progesterone therapy initiation and schedule a second ultrasound for six-months after progesterone initiation (+/- 7 days).

The second ultrasound will be performed after 6 months of progesterone therapy. Radiology technicians-blinded to the treatment groups-will measure the endometrial lining while performing the ultrasound. The radiologist will confirm and transcribe these results in an ultrasound report in the participant's medical record. A single reviewer board certified in gynecology will confirm endometrial stripe measurements as documented by the radiologist (+/-0.2cm). If there is discordance between measurements, a third gynecologist will review the ultrasound and make the final assessment of endometrial stripe thickness to ensure consistency with measurements.

In addition to ultrasound data, the study team will collect participant self-report data. Participants will be asked to complete brief REDCap questionaries at 3- and 6 months after progesterone initiation. Questionnaires will query participants' demographic characteristics, bleeding patterns, side effects, satisfaction, and adherence to the medication. For participants in the micronized progesterone treatment arm, they will be asked to save and bring their pill bottles at the 6 month visit (a total of two pill bottles); the study team will perform pill counts or patients will upload a picture to their file of their remaining pills to assess compliance.

All data will be stored securely in the REDCap database. Participants will be compensated a total of $50 in gift cards for their participation in the study, per table below.

D. Description, Risks and Justification of Procedures and Data Collection Tools:

This study involves minimal risks to participants. There is a potential risk for loss of privacy and confidentiality. Every reasonable effort will be made to protect participant information. All data will be stored in a secure, HIPAA-compliant REDCap database. Only authorized users that have completed the appropriate trainings will be granted access to the REDCap project. Data containing patient identifiers (MRNs, service dates) will only be stored in the project database for organizational purposes and will not be exported into the final data set used for analysis. Only de-identified data will be analyzed reported in future publications.

In terms of safety of ultrasound in this patient population, pelvic ultrasounds are routinely used in the field of pediatric and adolescent gynecology and is the preferred imaging modality to identify pelvic structures. Ultrasounds themselves are safe with no ionizing radiation or risk to surrounding structures with use of ultrasound itself. A trans-abdominal approach to pelvic ultrasound is often used in young adolescent patients due to its less invasive nature. However, the gold standard for identifying pelvic structures (in particular, the endometrial lining) is use of a transvaginal ultrasound probe. The transvaginal ultrasound probe can be painful and invasive for patients, especially those who have never used tampons or are not sexually active. Therefore, we will give our patients the option for the ultrasound approach with which they are most comfortable.

Data Safety and Monitoring Plan Definitions

1. Adverse Events (AE): An AE is defined as any unfavorable medical occurrence in a human subject, temporarily associated with the subject's participation in the research study, regardless of relationship to research participation. For the purposes of this study, AEs include any events that occur because of a study procedure (i.e., transabdominal ultrasound). As this study observes the effects of a progesterone therapy selected by the participant as part of their standard of care, events that occur because of the progesterone are monitored and managed by the participant's clinical team.
2. Serious Adverse Events (SAE): SAEs are defined as any adverse event associated with a subject's participation in research that is life threatening, requires inpatient hospitalization, results in a significant disability, results in a fetal anomaly, or results in death.
3. Unanticipated Problems (UPs): UPs can include AE/SAEs that are unanticipated events related directly to participant safety or protocol deviations that put participant privacy or confidentiality at risk. These UPs are unexpected, related to participation in research, and place participants at a greater risk of harm than was previously known or recognized.
4. Protocol Deviations: A generally unplanned deviation from the protocol that is not implemented or intended as a systematic change to the study protocol. This may include enrollment of an ineligible participant and missed study visits (i.e., ultrasounds).

Assessments The study PI will collect all AEs from the date informed consent is signed until the final study visit. All AEs, SAEs, UPs, and protocol deviations will be captured on the appropriate case report form (CRF). Information collected will include event description; time of onset; assessment of seriousness, severity, relationship to study procedures, expectedness, medical care received, outcomes of event, and time of resolution.

Reporting All AEs will be reported to COMIRB in aggregate as part of the continuing review. All SAEs will be reported to COMIRB within 48 hours of the Study PI becoming aware of the event. If UPs occur during the study, they will be reported to COMIRB within 48 hours of the Study PI becoming aware of the event, further, protocol deviations that influence participant safety will be reported to COMIRB within 48 hours of PI awareness.

Monitoring The primary investigator is responsible for ensuring participants' safety throughout this study and for reporting AEs, SAEs, and UPs to COMIRB according to the timeframes listed above. The PI will review procedures for maintaining the confidentiality of the data, the quality of data collection, data management, and analyses on a semiannual basis.

Data Analysis Plan:

Endometrial lining thickness and character will be collected via formal ultrasound report by the radiologist. We will report descriptive statistics for all outcomes of interest, including continuous endometrial thickness, and categorical descriptors provided in the ultrasound report. Descriptive statistics will be presented for factors that may influence patients' estrogen levels and response to estrogen replacement including etiology of the patient's ovarian failure, current estrogen therapy formulations and doses, BMI, age, and treatment group. Due to the potential for self-selection bias, we will compare the descriptive characteristics of the baseline endometrial lining by treatment group to investigate potential differences that may exist prior to treatment that may influence the primary outcome.

We will report descriptive statistics for each of the outcomes of interest. For categorical variables, we will report count and proportion, and for continuous variables we will report mean, SD, median, and IQR. We will descriptively compare the outcomes between the two treatment groups. All data will be collected and managed using REDCap.

The change in endometrial thickness will be calculated by comparing ultrasound findings at 6 months compared to patients' baseline ultrasound. Descriptive statistics will be reported for change in endometrial thickness by group, including mean, standard deviation (SD), range, median, and interquartile range (IQR). We will assess the distribution of the outcome using graphical methods, and we will use a parametric or non-parametric test as appropriate. We will test for a significant difference in the mean change between groups using a two-sample t-test in the case of a parametric distribution, and a Mann-Whitney-Wilcoxon test in the case of a non-parametric distribution. Data analysis will be conducted using R4.1.1.

Power and Sample Size We will enroll 34 participants, with at least 10 in each group (daily oral micronized progesterone or etonogestrel implant) and, ideally, 17 in each group. The study team will carefully track the number of participants enrolled in each group. When 17 are achieved in one group, study enrollment into that group will close. The study team will continue to present the study to eligible individuals and track the number interested in the closed treatment arm. Those individuals will be informed that they are not eligible for participation and thanked for their time. A sample of 34 participants who complete the study will achieve 80% power to detect a mean difference of 1 unit (mm) with a standard deviation of 1 unit. This sample size will also provide sufficient data to estimate a mean and standard deviation in the two study groups, to help power a non-inferiority design in a larger study.

Summarize Knowledge to be Gained:

This is a prospective study at a large tertiary center with high rates of hormone replacement therapy prescription for adolescent and young adult females. The information gained through this study is to generate pilot data for a larger, multisite study. Our long-term goals are to evaluate endometrial thickness based on imaging findings and to correlate these findings histologically via endometrial biopsies.

The proposed interventions of oral progesterone and the etonogestrel implant are safe medications that are accessible and already used widely in this patient population. We know that a trans-abdominal pelvic ultrasound to assess endometrial stripe thickness is a safe, non-invasive, and inexpensive method to evaluate endometrial thickness. To our knowledge, this is the first study to assess the effects of continuous progestin therapy in the pre-menopausal patient population regarding endometrial protection. Further, it is the first study of its kind to evaluate the effects of continuous etonogestrel and the etonogestrel implant on endometrial thickening in any patient population.

Currently there is a lack of research on the effect of the etonogestrel implant on endometrial thickness among patients using estrogen replacement therapy. Additionally, there is no available data regarding continuous oral micronized progesterone for the use of endometrial protection among patients using hormone replacement therapy who are not post-menopausal. This initial pilot data will provide a basis on how to best perform and power a future non-inferiority study.

There is also a lack of research on bleeding patterns among AYA female patients on combination hormone replacement therapy. Bothersome bleeding is one of the most common reasons for non-compliance and discontinuation of HRT in clinical practice; thus, it is prudent to determine differences in bleeding profiles between progesterone therapies. Additionally, we know that patients who are amenorrheic may have a different character and thickness to their endometrial stripe on ultrasound compared to those who are not amenorrheic. Gathering this information will allow us to stratify our analysis of endometrial thickness based on patients' reported bleeding patterns.

Studies that have evaluated and characterized endometrial stripe thickness via ultrasound have focused on post-menopausal populations. There is no standard endometrial thickness in the pre-menopausal population that is deemed to be pathologic or that requires intervention. Characterizing the endometrial lining on estrogen replacement therapy prior to initiating progesterone will both provide novel information about ultrasound findings of the endometrial lining in this patient population. It will also offer a baseline assessment by which to measure a change in endometrial thickness over the course of six months of progesterone therapy between study groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-25 years at baseline
* Female assigned at birth, with uterus
* Diagnosis of primary ovarian insufficiency or hypogonadotropic hypogonadism, requiring estrogen replacement therapy
* Receiving estradiol therapy-oral (1-2mg) or transdermal (0.05-0.1mg)-for at least 3 months
* Never used progesterone therapy or discontinued progesterone therapy at least 90-days prior to enrollment
* Consents to initiating progesterone therapy

Exclusion Criteria:

* Uterine abnormality (e.g., Müllerian Anomaly, uterine fibroids)
* Inability to characterize the endometrial lining on ultrasound
* History of chemotherapy or radiation therapy
* Inability to complete study questionnaire

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes 34 adolescent young adult individuals assigned female at birth, ages 12-25 years with a uterus in place, presenting to Children's Hospital Colorado-affiliated clinics: Pediatric and Adolescent Gynecology Clinic, Endocrine Clinic, Oncofertility Clinic, and Multidisciplinary Turner's Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in endometrial thickness after 6 months of progesterone therapy | 6 months
  Measure the mean change and variability in endometrial thickness (mm) in AYA treated for 6 months with either the etonogestrel implant or continuous oral progesterone via transabdominal pelvic ultrasound.

SECONDARY OUTCOMES:
Measure the mean endometrial thickness on estrogen replacement therapy | At least 3 months on estrogen replacement therapy
  Measure the mean endometrial thickness (mm) in AYA on estrogen hormone replacement therapy before initiation of progesterone therapy via transabdominal pelvic ultrasound.

OTHER OUTCOMES:
Satisfaction of progesterone replacement therapy | 6 months
  Assess overall satisfaction in AYA treated for 6 months with either the etonogestrel implant or continuous progesterone. This will be assessed via qualitative survey measures (10 point Likert scale).
Bleeding patterns on progesterone replacement therapy | 6 months
  Assess satisfaction with bleeding patterns in AYA treated for 6 months with either the etonogestrel implant or continuous progesterone. This will be assessed via qualitative survey measures (10 point Likert scale) and description of bleeding pattern (free response)
Side effects of progesterone replacement therapy | 6 months
  Assess side effects in AYA treated for 6 months with either the etonogestrel implant or continuous progesterone. This will be assessed via qualitative survey measures (free response).
Adherence to progesterone replacement therapy | 6 months
  Assess adherence in AYA treated for 6 months with either the etonogestrel implant or continuous progesterone. This will be assessed via qualitative survey in which participants will self report days of missed doses.
Rate of enrollment and attrition | 12 months
  Measure rate of patient enrollment (eg. non-eligible versus eligible, declined, enrolled) and attrition (eg. withdrawal from study, drop out, non-compliance) in each study arm within 12 months.
Number of patients willing to be randomized in future trial | 12 months
  Enrolled patients will indicate via survey their willingness to enroll in a future randomized control trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soontrapa N, Rattanachaiyanont M, Warnnissorn M, Wongwananuruk T, Indhavivadhana S, Tanmahasamut P, Techatraisak K, Angsuwathana S. The effectiveness of desogestrel for endometrial protection in women with abnormal uterine bleeding-ovulatory dysfunction: a non-inferiority randomized controlled trial. Sci Rep. 2022 Jan 31;12(1):1662. doi: 10.1038/s41598-022-05578-0. PMID 35102226
- [Background] Stanczyk FZ, Hapgood JP, Winer S, Mishell DR Jr. Progestogens used in postmenopausal hormone therapy: differences in their pharmacological properties, intracellular actions, and clinical effects. Endocr Rev. 2013 Apr;34(2):171-208. doi: 10.1210/er.2012-1008. Epub 2012 Dec 13. PMID 23238854
- [Background] Berlan ED, Richards MJ, Vieira CS, Creinin MD, Kaunitz AM, Fraser IS, Edelman A, Mansour D. Best Practices for Counseling Adolescents about the Etonogestrel Implant. J Pediatr Adolesc Gynecol. 2020 Oct;33(5):448-454. doi: 10.1016/j.jpag.2020.06.022. Epub 2020 Jul 2. PMID 32621879
- [Background] Stuenkel CA, Davis SR, Gompel A, Lumsden MA, Murad MH, Pinkerton JV, Santen RJ. Treatment of Symptoms of the Menopause: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2015 Nov;100(11):3975-4011. doi: 10.1210/jc.2015-2236. Epub 2015 Oct 7. PMID 26444994
- [Background] Committee Opinion No. 698: Hormone Therapy in Primary Ovarian Insufficiency. Obstet Gynecol. 2017 May;129(5):e134-e141. doi: 10.1097/AOG.0000000000002044. PMID 28426619
- [Background] Goncalves CR, Vasconcellos AS, Rodrigues TR, Comin FV, Reis FM. Hormone therapy in women with premature ovarian insufficiency: a systematic review and meta-analysis. Reprod Biomed Online. 2022 Jun;44(6):1143-1157. doi: 10.1016/j.rbmo.2022.02.006. Epub 2022 Feb 15. PMID 35461762
- [Background] Committee Opinion No. 698 Summary: Hormone Therapy in Primary Ovarian Insufficiency. Obstet Gynecol. 2017 May;129(5):963-964. doi: 10.1097/AOG.0000000000002040. PMID 28426614
- [Background] Effects of hormone replacement therapy on endometrial histology in postmenopausal women. The Postmenopausal Estrogen/Progestin Interventions (PEPI) Trial. The Writing Group for the PEPI Trial. JAMA. 1996 Feb 7;275(5):370-5. doi: 10.1001/jama.1996.03530290040035. PMID 8569016
- [Background] Lobo RA, Archer DF, Kagan R, Kaunitz AM, Constantine GD, Pickar JH, Graham S, Bernick B, Mirkin S. A 17beta-Estradiol-Progesterone Oral Capsule for Vasomotor Symptoms in Postmenopausal Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):161-170. doi: 10.1097/AOG.0000000000002645. PMID 29889748
- [Background] Mueck AO, Romer T. Choice of progestogen for endometrial protection in combination with transdermal estradiol in menopausal women. Horm Mol Biol Clin Investig. 2018 Jul 31;37(2). doi: 10.1515/hmbci-2018-0033. PMID 30063464
- [Background] Popat VB, Calis KA, Kalantaridou SN, Vanderhoof VH, Koziol D, Troendle JF, Reynolds JC, Nelson LM. Bone mineral density in young women with primary ovarian insufficiency: results of a three-year randomized controlled trial of physiological transdermal estradiol and testosterone replacement. J Clin Endocrinol Metab. 2014 Sep;99(9):3418-26. doi: 10.1210/jc.2013-4145. Epub 2014 Jun 6. PMID 24905063
- [Background] Sullivan SD, Sarrel PM, Nelson LM. Hormone replacement therapy in young women with primary ovarian insufficiency and early menopause. Fertil Steril. 2016 Dec;106(7):1588-1599. doi: 10.1016/j.fertnstert.2016.09.046. PMID 27912889
- [Background] Armeni E, Paschou SA, Goulis DG, Lambrinoudaki I. Hormone therapy regimens for managing the menopause and premature ovarian insufficiency. Best Pract Res Clin Endocrinol Metab. 2021 Dec;35(6):101561. doi: 10.1016/j.beem.2021.101561. Epub 2021 Jun 30. PMID 34274232
- [Background] "The 2022 Hormone Therapy Position Statement of The North American Menopause Society" Advisory Panel. The 2022 hormone therapy position statement of The North American Menopause Society. Menopause. 2022 Jul 1;29(7):767-794. doi: 10.1097/GME.0000000000002028. PMID 35797481
- [Background] Divasta AD, Gordon CM. Hormone replacement therapy and the adolescent. Curr Opin Obstet Gynecol. 2010 Oct;22(5):363-8. doi: 10.1097/GCO.0b013e32833e4a35. PMID 20724926
- [Background] Cattoni A, Parissone F, Porcari I, Molinari S, Masera N, Franchi M, Cesaro S, Gaudino R, Passoni P, Balduzzi A. Hormonal replacement therapy in adolescents and young women with chemo- or radio-induced premature ovarian insufficiency: Practical recommendations. Blood Rev. 2021 Jan;45:100730. doi: 10.1016/j.blre.2020.100730. Epub 2020 Jul 4. PMID 32654893